CLINICAL TRIAL: NCT03427099
Title: The Effect of a Developed Perioperative Rehabilitation Pathway Following Lumbar Arthrodesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other); UHasselt (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KU/UZ Leuven S60109 - 3
Record Dates: First submitted 2018-01-26; First posted 2018-02-09 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Physical Disability; Low Back Pain, Recurrent; Surgery
MeSH Terms: conditions — Low Back Pain | interventions — Rehabilitation; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): usual care
  Interventions: Behavioral: Control group
- Intervention group (Experimental): Rehabilitation with a biopsychosocial focus
  Interventions: Behavioral: Rehabilitation with a biopsychosocial focus

INTERVENTIONS:
Behavioral: Rehabilitation with a biopsychosocial focus — Rehabilitation with a biopsychosocial focus
  Arms: Intervention group
Behavioral: Control group — usual care
  Arms: Control group

SUMMARY:
To compare the current rehabilitation pathway with the implementation of a newly developed rehabilitation pathway for patients with a single and double level lumbar arthrodesis.

DETAILED DESCRIPTION:
This involves a prospective interventional study with a one year follow-up. The investigators will compare the outcomes of the current rehabilitation pathway with a newly developed (based on systematic review and delphi study) rehabilitation pathway for patients with a single and double level lumbar arthrodesis. The usual care group (n= 30) will be compared with the intervention group (n= 30).

ELIGIBILITY:
Inclusion Criteria:

* Lumbar single and double level arthrodesis
* Signed informed consent
* Posterior Lumbar interbody fusion (PLIF), Posterolateral lumbar fusion (PLF) and Transforaminal lumbar interbody fusion (TLIF)

Exclusion Criteria:

* Previous arthrodesis in the lumbar spine
* Musculoskeletal disorders which interfere with functional outcome, f.e. severe lower limb problems not related to the lumbar surgery
* Presence of one of the following pathologies:Parkinson Multiple sclerose (MS), Cerebral vascular accident (CVA), Peripheral neuropathies, Circulatory disorders, Gout, Rheumatoid disorders, Neoplasia, Septic arthritis, Pregnancy, Vestibular disorder, Infectious diseases
* Accident at work or lawsuit
* Low cognition
* Not able to speak Dutch

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | Postoperative: 1 week
  questionnaire measuring disability related to low back pain
Oswestry Disability Index (ODI) | Postoperative: 6 weeks
  questionnaire measuring disability related to low back pain
Oswestry Disability Index (ODI) | Postoperative: 3 months
  questionnaire measuring disability related to low back pain
Oswestry Disability Index (ODI) | Postoperative: 6 months
  questionnaire measuring disability related to low back pain
Oswestry Disability Index (ODI) | Postoperative: 1 year
  questionnaire measuring disability related to low back pain

SECONDARY OUTCOMES:
Numeric Rating scale (NRS) | Postoperative: 1 week, 6 weeks, 3 months, 6 months, 1 year
  Severity of low back pain will be scored by the Numerical Rating Scale (NRS) from zero ('no pain') to ten ('worst pain imaginable') (Jensen, M.P., Karoly, P., Braver, S. (1986). The measurement of clinical pain intensity: a comparison of six methods. Pain 27, 117-126.)
Tampa scale for Kinesiophobia (TSK) | Postoperative: 1 week, 6 weeks, 3 months, 6 months, 1 year
  The Tampa Scale for Kinesiophobia (TSK), which ranges from 17 ('low') to 68 ('high'), was completed to identify fear of (re)injury following movements or activities in the participants with low back pain (Kori, K.S., Miller, R.P., Todd, D.D. (1990). Kinesiophobia: A new view of chronic pain behaviour. Pain 3, 35-43.)
Pain Catastrophizing scale (PCS) | Postoperative: 1 week, 6 weeks, 3 months, 6 months, 1 year
  People are asked to indicate the degree to which they have the above thoughts and feelings when they are experiencing pain using the 0 (not at all) to 4 (all the time) scale. A total score is yielded (ranging from 0-52), along with three subscale scores assessing rumination, magnification and helplessness.
Depression Anxiety stress scale (DASS) | Postoperative: 1 week, 6 weeks, 3 months, 6 months, 1 year
  A higher score on the DASS indicates greater severity or frequency of negative emotional symptoms, ranging from 0-126.
EuroQol five dimensions questionnaire (EQ-5D) | Postoperative: 1 week, 6 weeks, 3 months, 6 months, 1 year
  questionnaire measuring general health
Sit-to-stand | Postoperative: 1 week, 6 weeks, 3 months, 6 months, 1 year
  time to perform 5 times sit-to-stand-to-sit
Patient Specific Functional Scale (PSFS) | Postoperative: 1 week, 6 weeks, 3 months, 6 months, 1 year
  The PSFS is a questionnaire measuring disability related to low back pain. The Scale is developed by "Stratford, P., Gill, C., Westaway, M., & Binkley, J. (1995). Assessing disability and change on individual patients: a report of a patient specific measure. Physiotherapy Canada, 47, 258-263." Three to five activities are scored on a Visual Analogue Scale (VAS) from 0 ('not able to perform activity') to 10 ('can perform activity without any problems'). Lower scores indicate a worse outcome on function. The total score is the sum of the VAS scores of the 3 to 5 activities.
Return-to-work | Postoperative: 1 week, 6 weeks, 3 months, 6 months, 1 year
  questionnaire on work resumption

CONTACTS AND LOCATIONS:
Overall Officials: Bart Depreitere, PhD, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Thijs Swinnen, MSc, PT, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Tinne Thys, MSc, PT, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Wim Dankaerts, PhD, PT, Principal Investigator — KU Leuven; Simon Brumagne, PhD, PT, Principal Investigator — KU Leuven; Peter Van Wambeke, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Lieven Moke, PhD, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Sebastiaan Schelfaut, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Ann Spriet, MSc, PT, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Lotte Janssens, PhD, PT, Principal Investigator — Hasselt University
Locations (1):
- UZ/KU Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided